CLINICAL TRIAL: NCT03734289
Title: Improving Family Quality of Life Through Training to Reduce Care-Resistant Behaviors by People With Alzheimer Dementia and Traumatic Brain Injury (NeuroNS) Study
Brief Title: Improving Family Quality of Life Through Training to Reduce Care-Resistant Behaviors by People With AD and TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Geldmacher, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-160819003; W81XWH-16-1-0527 (Other Grant/Funding Number: US Dept of Defense); CDMRP-AZ150084 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2018-10-09; First posted 2018-11-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Traumatic Brain Injury
MeSH Terms: conditions — Dementia; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Caregivers will be randomized in a 1:1 ratio for immediate intervention vs. a 6 week delayed intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Coaching (Active Comparator): Immediately following randomization, online coaching sessions will occur weekly for 6 weeks. Web-based courses containing instructional materials that deal with preventing and reducing care resistant behavior (CRB) within intimate care (dressing, bathing, toileting) and treatment regimens (medication, therapeutic activities) after the initial study visit. The NeuroNS-Care intervention is an innovative distance-learning , internet based, family caregiver coaching program; one for the caregivers of persons with dementia and one for the caregivers of persons recovering from TBI. It will be delivered using Instructure's Canvas™ web-based platform.
  Interventions: Behavioral: Caregiver Coaching
- Delayed Coaching (Active Comparator): 6 weeks following the initial visit, online coaching sessions will occur weekly for 6 weeks. Web-based courses containing instructional materials that deal with preventing and reducing care resistant behavior (CRB) within intimate care (dressing, bathing, toileting) and treatment regimens (medication, therapeutic activities) after the initial study visit. The NeuroNS-Care intervention is an innovative distance-learning , internet based, family caregiver coaching program; one for the caregivers of persons with dementia and one for the caregivers of persons recovering from TBI. It will be delivered using Instructure's Canvas™ web-based platform.
  Interventions: Behavioral: Caregiver Coaching

INTERVENTIONS:
Behavioral: Caregiver Coaching — Online coaching sessions will occur weekly for 6 weeks. Web-based courses containing instructional materials that deal with preventing and reducing care resistant behavior (CRB) within intimate care (dressing, bathing, toileting) and treatment regimens (medication, therapeutic activities) after the initial study visit. The NeuroNS-Care intervention is an innovative distance-learning , internet based, family caregiver coaching program; one for the caregivers of persons with dementia and one for the caregivers of persons recovering from TBI. It will be delivered using Instructure's Canvas™ web-based platform.

SUMMARY:
To reduce care resistant behaviors (CRB) among people with dementia residing in nursing homes, to a distance-learning education, training, and coaching program for family caregivers of people with dementia or TBI; assess the efficacy of the intervention for reducing frequency or severity of CRB-triggered symptoms of agitation, aggression, and irritability; assess the efficacy of the intervention for improving quality of life of patients, caregivers, and families; and determine how patient and caregiver characteristics influence the effectiveness of the intervention.

5. Evaluate how the intervention affects the health care costs of people with dementia or TBI.

DETAILED DESCRIPTION:
To address the previously unanswered question of whether theoretically-driven caregiver education and coaching in nonpharmacologic approaches to reduce care resistant behaviors as a trigger of behavioral and psychiatric symptoms of dementia (BPSD) and neuropsychiatric symptoms after Traumatic Brain Injury (NPTBI) will improve caregiver burden, quality of life (QOL), and related outcomes of patients with these conditions and their family members. The intervention of interest is the Neurobehavioral Non-Pharmacologic Supportive Strategies for Family Caregivers of Persons with Dementia or TBI (NeuroNS-Care). Behavioral symptoms in dementia and following TBI vary considerably over time, with a tendency toward spontaneous regression to the mean. Additionally, caregivers often develop idiosyncratic strategies in response to adverse behaviors that might be either adaptive or maladaptive. In order to separate the effects of time alone from the effects of the coaching intervention, one group will be randomized to delayed intervention following a 6 week wait time. This will allow the investigative team the opportunity to compare the natural history of the outcome variables in an "untrained" portion of the sample to the effects of training over a similar time period.

ELIGIBILITY:
50 participants with possible or probable Alzheimer's disease dementia (of all severity stages) as defined by the NIA-Alzheimer's Association 2011 criteria will be enrolled, along with a family (i.e., unpaid) caregiver. A second cohort of 25 participants who have sustained moderate to severe TBI as diagnosed by UAB-TBIMS standards (generally Glasgow Coma Scale score of 12 or less at admission, cranial imaging with evidence of acute intracranial trauma, and/or post-traumatic amnesia duration of greater than 24 hours) ≥6 months prior to study entry (and their caregivers) will be enrolled.

Entry is dependent on caregiver ratings on at least one of three behavioral domains of the Neuropsychiatric Inventory (NPI): 1) Agitation/Aggression, 2) Disinhibition, 3) Irritability /Lability. Based on standard scoring of the NPI, the caregiver must report all of these for at least one domain:

* Frequency of "Often" (several times per week but less than every day) or more,
* Severity of "Moderate" (stressful and upsetting; may require specific management) or higher
* Distress of "Moderate" (fairly distressing, not always easy to cope with) or higher

The caregiver must also report that the adverse behavior is triggered by resistance to care-related activities, e.g., bathing, taking medications, attending health-care appointments, etc.

Additional inclusion criteria.

* Age ranges AD: ≥ 50 years; TBI ≥ 19; Caregiver ≥18
* Sex distribution: both men and women.
* Race: any.
* Health: generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane). Vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures, or participants who per clinician criteria are deemed eligible to participate in the study. .
* Cognitive function and spoken/written English language skills sufficient to provide valid results on neuropsychological testing, or participants who per clinician criteria are deemed eligible to participate in the study.
* Concomitant medications: Subjects may be on stable doses of any psycho-active agents for ≥30 days prior to screening and randomization.
* Caregiver: unpaid person who provides support or supervision for at least 1 instrumental activity of daily living for the affected person, with direct contact averaging ≥5 of every 7 days, and ≥21 hours weekly.
* Access to high-speed/broad band internet service through home computer capable of operating "Go-to-Meeting" or equivalent conferencing software.

Exclusion criteria.

* Absence of a reliable caregiver who is willing to participate and comply with protocol responsibilities (described below).
* Evidence of other psychiatric/neurologic disorders sufficient to be the primary source of cognitive impairment (i.e., stroke, idiopathic Parkinson's disease, schizophrenia, bipolar or unipolar depression, seizure disorder).
* Psychotic features (delusions or hallucinations) not adequately treated or not on stable medical therapy for these conditions 30 days prior to enrollment.
* Current or recent (within the past 2 years) history of alcoholism or drug misuse.
* Subject and/or caregivers who are unwilling or unable to fulfill the requirements of the study.
* Any condition which would make the subject or the caregiver, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Zarit Burden Interview | Change from baseline to 6-month follow-up
  A measure of caregiver burden

SECONDARY OUTCOMES:
Change in Dementia Quality of Life (DEMQOL/DEMQOL proxy) | Change from baseline through 6-month follow-up
  Measures of quality of life for the person with dementia
Change in Neuropsychiatric Inventory | Change from baseline through 6-month follow-up
  Measure of behavioral symptomsand caregiver distress
Change in Family Quality of Life (Dementia or TBI versions) | Change from baseline through 6-month follow-up
  Measures of family function and family-based quality of life
Change in Connor-Davidson Resilience Scale (CD-RISC) | Change from baseline through 6-month follow-up
  Measure of caregiver resilience

CONTACTS AND LOCATIONS:
Overall Officials: David Geldmacher, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States